CLINICAL TRIAL: NCT07349212
Title: A First-in-Human, Ascending Dose, Open-label, Multicenter Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of UKK-0018 in Peanut Allergic Individuals
Brief Title: UKK-0018 is an Immunotherapeutic for Treatment of Peanut Allergies
Acronym: UKK-0018
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ukko Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKKO-18-101-ANZ
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Peanut-Induced Anaphylaxis; Peanut Allergy
Keywords: peanut; peanut allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: This is a first-in-human, open-label, multicenter study that will be conducted in adult participants (ages 18-55, inclusive) with peanut allergy in sequential cohorts evaluating dose levels and intervals (collectively called 'dose regimen').
  Based on emerging data an optional dose expansion cohort may be added, at a dose regimen to be determined.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UKK-0018 (Experimental): UKK0018 is an immunotherapeutic for the treatment of peanut allergies
  Interventions: Biological: UKK-0018

INTERVENTIONS:
Biological: UKK-0018 — UKK0018 is an immunotherapeutic treatment of peanut allergies

SUMMARY:
This study will test a new investigational treatment called UKK-0018. UKK-0018 is an immunotherapeutic for the treatment of peanut allergies. The treatment is given by injection and is designed to train the immune system to tolerate peanut exposure over time.

DETAILED DESCRIPTION:
The study will assess how safe and well tolerated UKK-0018 is in people with known peanut allergy, and whether it can reduce the risk of allergic symptoms following exposure to peanut proteins.

This is a first-in-human, open-label, multicenter study that will be conducted in adult participants with peanut allergy evaluating dose levels and regimens. It is anticipated that UKK-0018 can help retrain the immune system over time to respond safely to peanut proteins in case of accidental exposures. The modifications which reduce binding to IgE antibodies are anticipated to reduce risk of serious allergic reactions compared to standard of care.

Based on emerging data an optional dose expansion cohort may be added. An optional dose expansion cohort may be added if supported by emerging data. The study is comprised of a screening period, intervention period, and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-55 years old
* documented history of physician-diagnosed peanut allergy
* positive skin prick test (SPT)
* screening DBPCFC peanut protein
* contraception use should be consistent with local regulations
* capable of providing signed written informed consent

Exclusion Criteria:

* asthma based on NHLBI
* uncontrolled cardiovascular disease
* chronic disease history
* exacerbation of dermatological conditions
* life threatening episodes of anaphylaxis
* active infections
* poor physical or blood chemistry
* immunodeficiency, bleeding disorders, malignancies
* hypersensitivities to epinephrine, inactive ingredients in therapy
* pregnant or breast feeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of repeated dosing of UKK-0018 administered IM of solicited local and systemic adverse reactions | 7 days after each injection
  Numbers and percentages of participants with solicited local and systemic adverse reactions
To assess the safety and tolerability of repeated dosing of UKK-0018 administered IM of unsolicited adverse events | 28 days after each injection
  Numbers and percentages of participants with unsolicited adverse events (AEs)
To assess the safety and tolerability of repeated dosing of UKK-0018 administered IM of medically-attended adverse events (MAAEs | 30 weeks after first injection
  Numbers and percentages of participants with medically-attended adverse events (MAAEs)
To assess the safety and tolerability of repeated dosing of UKK-0018 administered IM of adverse events of special interest (AESI) | 30 weeks after first injection
  Numbers and percentages of participants with adverse events of special interest (AESI)
To assess the safety and tolerability of repeated dosing of UKK-0018 administered IM of serious adverse events (SAE) | 30 weeks after first injection
  Numbers and percentages of participants with serious adverse events (SAE)

SECONDARY OUTCOMES:
To assess the preliminary efficacy of repeated dosing of UKK-0018 administered IM in participants with peanut allergy | at 24 weeks post last treatment
  The number of participants able to increase their tolerated dose (eg, no more than mild dose-limiting symptoms) of peanut protein at least 10-fold in the exit double-blind placebo-controlled food challenge (DBPCFC) compared to the screening DBPCFC.
To assess the preliminary efficacy of repeated IM dosing of UKK-0018 in participants with peanut allergy | at 24 weeks post treatment
  The number of participants able to ingest ≥ 600 mg of peanut protein in a DBPCFC
To assess the effect of dose regimen on immunogenicity and biomarkers following repeated IM dosing of UKK-0018 | up to 30 weeks
  Change from baseline in immunogenicity markers measured by geometric mean ratios (GMRs) and 95% confidence intervals (CIs) at prespecified time points up to study completion

CONTACTS AND LOCATIONS:
Locations (2):
- The Royal Melbourne Hospital, Fitzroy, Victoria, Australia
- Pacific Clinical Research Network, Auckland, New Zealand